CLINICAL TRIAL: NCT02259114
Title: A Phase IB Trial With OTX015/MK-8628, a Small Molecule Inhibitor of the Bromodomain and Extra-Terminal (BET) Proteins, in Patients With Selected Advanced Solid Tumors
Brief Title: A Dose-Finding Study of Birabresib (MK-8628), a Small Molecule Inhibitor of the Bromodomain and Extra-Terminal (BET) Proteins, in Adults With Selected Advanced Solid Tumors (MK-8628-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncoethix GmbH, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8628-003; OTX015_108 (Other: OncoEthix); 2014-002680-15 (EudraCT Number); MK-8628-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: NUT Midline Carcinoma; Triple Negative Breast Cancer; Non-small Cell Lung Cancer With Rearranged ALK Gene/Fusion Protein or KRAS Mutation; Castrate-resistant Prostate Cancer; CRPC; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continuous Dosing Regimen (Experimental): Participants receive birabresib capsules once daily in a fasted state in the morning on Days 1-21 of each 21-day cycle. Starting dose for dose escalation is 80 mg.
  Interventions: Drug: Birabresib
- Days 1-7 Dosing Regimen (Experimental): Participants receive birabresib capsules once daily in a fasted state in the morning on Days 1-7 of each 21-day cycle. Starting dose for dose escalation is 100 mg.
  Interventions: Drug: Birabresib

INTERVENTIONS:
Drug: Birabresib — Birabresib 10, 20 and/or 40 mg oral capsules
  Other Names: OTX105; MK-8628

SUMMARY:
Open-label, phase I, non-randomized, multicentric study of single-agent birabresib (MK-8628) (formerly known as OTX015) administered according to two distinct regimens to participants with selected advanced tumors.

The study will be performed in two parts.

Dose Escalation Part:

This step is designed to determine the maximum tolerated dose (MTD) in each of the two regimens, which will be evaluated in parallel. Participants will receive oral birabresib according to:

Continuous Dosing Regimen: continuous, once daily for 21 consecutive days (21-day cycles).

OR Days 1-7 Dosing Regimen: once daily on Days 1 to 7, repeated every 3 weeks (21-day cycles; 1 week ON/2 weeks OFF).

Participants will be sequentially assigned to Continuous Dosing Regimen or Days 1-7 Dosing Regimen according to the next available place and receive birabresib at escalating doses levels (DL). Cohorts of 3 participants will be treated, and an additional 3 participants will be treated at the first indication of dose-limiting toxicity (DLT). MTD assessment will be based on the tolerability observed during the first 21 days of treatment.

Expansion Part:

The efficacy of birabresib in each of the five indications (i.e., Bromodomain-Nuclear Protein in Testis [BRD-NUT] midline carcinoma, triple negative breast cancer [TNBC], non-small cell lung cancer [NSCLC] harboring a rearrangement Anaplastic Lymphoma Kinase [ALK] gene/fusion protein or Kirsten Ras [KRAS] mutation, castrate-resistant prostate cancer, and pancreatic ductal carcinoma) will be assessed in terms of response (Response Evaluation Criteria in Solid Tumors v1.1 [RECIST v1.1] or Prostate Cancer Clinical Trials Working Group 2 [PCWG2]) using a selected regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures and treatment;
2. Histologically or cytologically confirmed diagnosis of one of the following advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective, intolerable or inacceptable for the patient:

   * NUT midline carcinoma (ectopic expression of NUT protein as determined by immunohistochemistry (IHC) and/or detection of BRD-NUT gene translocation as determined by fluorescence In situ hybridization [FISH]);
   * Triple negative breast cancer defined according to American Society of Clinical Oncology (ASCO) recommendations (Hammond et al., 2010; Wolff et al., 2007);
   * Non-small cell lung cancer harboring a rearranged ALK gene/fusion protein (FISH or IHC) or KRAS mutation (as defined by any molecular analysis);
   * Castrate-resistant prostate cancer (CRPC);
   * Pancreatic ductal adenocarcinoma;
3. At least one measurable lesion as per RECIST version 1.1., except for CRPC participants who may be enrolled with objective evidence of disease as per PCWG2 criteria;
4. Age ≥18 years at the time of informed consent;
5. Life expectancy ≥3 months;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤1;
7. Adequate bone marrow reserve, renal and liver function:

   * Absolute neutrophil count ≥1.5 x10^9/L,
   * Platelet count ≥150 x10^9/L,
   * Hemoglobin ≥9 g/dL,
   * Creatinine clearance ≥30 mL/min calculated according to the Cockroft and Gault formula or Modification of Diet in Renal Disease (MDRD) formula for participants aged >65 years,
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) and total bilirubin ≤1.25 x ULN (in case of liver involvement, ALT/AST ≤5 x ULN and total bilirubin ≤2 x ULN will be allowed),
   * Serum albumin ≥2.8 g/dL,
   * International Normalized Ratio (INR) ≤1.5 x ULN or INR <3 for participants treated with antivitamin K;
8. An interval of ≥3 weeks since chemotherapy (≥6 weeks for nitrosoureas or mitomycin C), immunotherapy, hormone therapy or any other anticancer therapy or surgical intervention resection, or ≥3 half-lives for monoclonal antibodies, or ≥5 half-lives for other non-cytotoxic agents (whichever is longer);
9. CRPC participants must maintain ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue, antagonist or orchiectomy providing serum testosterone is <50 ng/dL (<1.7 nmol/L);
10. Participants receiving bisphosphonate or denosumab therapy must be on stable doses for at least 4 weeks before initiating study treatment.

Exclusion Criteria:

1. Inability to swallow oral medications or presence of a gastrointestinal disorder (e.g. malabsorption) deemed to jeopardize intestinal absorption of birabresib;
2. Persistent grade >1 clinically significant toxicities related to prior antineoplastic therapies (except for alopecia); stable sensory neuropathy ≤ grade 2 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.0 is accepted.
3. Known primary central nervous system (CNS) malignancy or CNS involvement;
4. History of prior or concomitant malignancies (other than excised non-melanoma skin cancer or cured in situ cervical carcinoma) within 3 years of study entry;
5. Other serious illness or medical conditions, such as active infection, unresolved bowel obstruction, or psychiatric disorders;
6. Known human immunodeficiency virus (HIV) positivity;
7. Participation in another clinical trial or treatment with any investigational drug within 30 days prior to study entry;
8. Other concomitant anticancer treatment;
9. Concomitant therapy with strong CYP3A4 interfering drugs;
10. Current use of anticoagulants (e.g. warfarin, heparin) at therapeutic levels within 7 days prior to the first dose of birabresib. Low-dose (prophylactic) low molecular weight heparin (LMWH) is permitted;
11. Pregnant or breast-feeding participants, and men and women with childbearing potential not using effective contraception while on study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Lewin J, Soria JC, Stathis A, Delord JP, Peters S, Awada A, Aftimos PG, Bekradda M, Rezai K, Zeng Z, Hussain A, Perez S, Siu LL, Massard C. Phase Ib Trial With Birabresib, a Small-Molecule Inhibitor of Bromodomain and Extraterminal Proteins, in Patients With Selected Advanced Solid Tumors. J Clin Oncol. 2018 Oct 20;36(30):3007-3014. doi: 10.1200/JCO.2018.78.2292. Epub 2018 May 7. PMID 29733771
- [Derived] Vazquez R, Riveiro ME, Astorgues-Xerri L, Odore E, Rezai K, Erba E, Panini N, Rinaldi A, Kwee I, Beltrame L, Bekradda M, Cvitkovic E, Bertoni F, Frapolli R, D'Incalci M. The bromodomain inhibitor OTX015 (MK-8628) exerts anti-tumor activity in triple-negative breast cancer models as single agent and in combination with everolimus. Oncotarget. 2017 Jan 31;8(5):7598-7613. doi: 10.18632/oncotarget.13814. PMID 27935867

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8628 Continuous Dosing Regimen 80 mg/Day: Participants received MK-8628 (formerly OTX015) capsules at a total daily dose of 80 mg/day once daily in a fasted state in the morning on Days 1-21 of each 21-day cycle.
- MK-8628 Continuous Dosing Regimen 100 mg/Day: Participants received MK-8628 capsules at a total daily dose of 100 mg/day once daily in a fasted state in the morning on Days 1-21 of each 21-day cycle.
- MK-8628 Days 1-7 Dosing Regimen 100 mg/Day: Participants received MK-8628 capsules at a total daily dose of 100 mg/day once daily in a fasted state in the morning on Days 1-7 of each 21-day cycle.
- MK-8628 Days 1-7 Dosing Regimen 120 mg/Day: Participants received MK-8628 capsules at a total daily dose of 120 mg/day once daily in a fasted state in the morning on Days 1-7 of each 21-day cycle.
- MK-8628 Days 1-7 Dosing Regimen 160 mg/Day: Participants received MK-8628 capsules at a total daily dose of 160 mg/day once daily in a fasted state in the morning on Days 1-7 of each 21-day cycle.
Period: Overall Study
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Started | 21 | 4 | 13 | 3 | 6
Treated | 20 (One participant was randomized but did not receive treatment due to a protocol violation.) | 4 | 13 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 21 | 4 | 13 | 3 | 6
Not completed — Progressive Disease | 14 | 2 | 10 | 2 | 5
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 1
Not completed — Death | 3 | 0 | 1 | 0 | 0
Not completed — Treatment Delay >2 wks: Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0
Not completed — Treatment Delay >2 wks: Toxicity | 1 | 1 | 0 | 0 | 0
Not completed — Not Treated | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all participants who received at least one dose of study treatment.
Groups:
- MK-8628 Continuous Dosing Regimen 80 mg/Day: Participants received MK-8628 capsules at a total daily dose of 80 mg/day once daily in a fasted state in the morning on Days 1-21 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day | Total
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (18.8) | 62.5 (13.5) | 64.3 (9.5) | 63.3 (9.3) | 58.5 (5.3) | 57.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 0 | 0 | 1 | 7
  Male | 15 | 3 | 13 | 3 | 5 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT) During Cycle 1
Description: A DLT was defined as any of the following toxicities that were considered by the investigator to be related to MK-8628: Hematologic toxicity: Grade 4 hematologic toxicity or febrile neutropenia, Grade 3 neutropenia with infection, Grade 3 thrombocytopenia with bleeding or lasting >7 days; Non-hematologic toxicity: Grade 3 or 4 non-hematologic toxicity (regardless of duration) unless it was not optimally managed with supportive care, Grade 3 or 4 laboratory abnormality, with or without symptoms, lasting >48 hours, Intolerable Grade 2 non-hematologic toxicity resulting in study drug discontinuation or delay >7 days with or without dose reduction, Designated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) liver test abnormalities; Treatment delay >2 weeks or dose reduction requirement for initiating Cycle 2.
Time Frame: Up to Cycle 1 Day 21 (Up to 21 days)
Population: The DLT Evaluable Population consisted of all participants who received ≥85% of the planned dose of study treatment (18 days for Continuous Dosing Regimens, or 6 days for Days 1-7 Dosing Regimens) or experienced a DLT during the first 21-day cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Participants | 4 | 2 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence associated with use of study treatment in humans, whether or not considered treatment related. The number of participants who experienced at least one AE is presented.
Time Frame: Up to approximately 17.5 months (Up to 30 days after last dose of study treatment)
Population: The Safety Population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Participants | 20 | 4 | 13 | 3 | 6

3. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 16.5 months
Population: The Safety Population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Participants | 5 | 3 | 2 | 0 | 1

4. Secondary Outcome: Best Overall Response as Assessed in Solid Tumors by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or in Castration-resistant Prostate Cancer (CRPC) by Prostate Cancer Clinical Trials Working Group (PCWG2) Response Criteria
Description: The best overall response was the best response recorded from the start of the study treatment until the end of treatment. RECIST 1.1 response categories included: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions; and Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to approximately 16.5 months
Population: The Efficacy Population consisted of all participants who received ≥2 complete cycles (6 weeks) of study treatment and underwent baseline assessment and 1 on-study tumor assessment, or who discontinued early due to disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 19 | 2 | 12 | 3 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 3 | 0 | 0 | 0 | 0
  Stable Disease | 12 | 0 | 7 | 1 | 5
  Progressive Disease | 4 | 1 | 5 | 2 | 1
  Not Evaluable | 0 | 1 | 0 | 0 | 0

5. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) of MK-8628
Description: Blood samples were obtained at specified time points for pharmacokinetic (PK) analysis of the observed Cmax of MK-8628. The observed Cmax of MK-8628 after administration is presented.
Time Frame: Cycle 1 Day1: Predose; 0.25, 1, 2, 3 and 7 hours postdose
Population: The Pharmacokinetics (PK) Population consisted of all participants who received MK-8628 on Cycle 1 Day 1 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
μg/L | 1466 (566) | 1867 (241) | 1514 (377) | 2052 (1130) | 2670 (741)

6. Secondary Outcome: Time to Cmax (Tmax) of MK-8628
Description: Blood samples were obtained at specified time points for PK analysis of the Tmax of MK-8628. The Tmax of MK-8628 after administration is presented.
Time Frame: Cycle 1 Day1: Predose; 0.25, 1, 2, 3 and 7 hours postdose
Population: The PK Population consisted of all participants who received MK-8628 on Cycle 1 Day 1 and had blood samples drawn for PK analyses.
Measure: Median (Standard Deviation); unit: Hours
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Hours | 2.0 (0.6) | 2.4 (0.5) | 2.9 (0.7) | 1.9 (0.6) | 2.5 (0.6)

7. Secondary Outcome: Area Under to Concentration-Time Curve From 0 to Infinity (AUC0-∞) of MK-8628
Description: Blood samples were obtained at specified time points for PK analysis of the AUC0-∞ of MK-8628. The AUC0-first is AUC0-∞ which is derived from the post-hoc estimate of CL/F from the population model. The AUC0-∞ of MK-8628 after administration is presented.
Time Frame: Cycle 1 Day1: Predose; 0.25, 1, 2, 3 and 7 hours postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg*h/L
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
μg*h/L | 12550 (4456) | 19130 (6543) | 12800 (3597) | 16210 (9551) | 27440 (10510)

8. Secondary Outcome: Volume of Distribution at Steady State (Vdss) of MK-8628
Description: Blood samples were obtained at specified time points for PK analysis of the Vdss of MK-8628. The Vdss of MK-8628 after administration is presented.
Time Frame: Cycle 1 Day1: Predose; 0.25, 1, 2, 3 and 7 hours postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Liters | 44.9 (13.4) | 44.3 (5.59) | 46.9 (9.2) | 44.0 (18.3) | 41.6 (15.1)

9. Secondary Outcome: Terminal Half-Life (t1/2) of MK-8628
Description: Blood samples were obtained at specified time points for PK analysis of the t1/2 of MK-8628. The t1/2 of MK-8628 after administration is presented.
Time Frame: Cycle 1 Day1: Predose; 0.25, 1, 2, 3 and 7 hours postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Hours | 4.53 (0.866) | 5.93 (2.46) | 3.97 (0.46) | 3.52 (0.593) | 3.99 (0.664)

10. Secondary Outcome: Total Plasma Clearance (CL) of MK-8628
Description: Blood samples were obtained at specified time points for PK analysis of the CL of MK-8628. The CL of MK-8628 after administration is presented.
Time Frame: Cycle 1 Day1: Predose; 0.25, 1, 2, 3 and 7 hours postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters/Hour
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
Number analyzed (Participants) | 20 | 4 | 13 | 3 | 6
Liters/Hour | 6.98 (1.98) | 5.69 (1.87) | 8.36 (2.16) | 8.97 (4.02) | 7.39 (2.76)

ADVERSE EVENTS:
Time Frame: Up to approximately 17.5 months (Up to 30 days after last dose of study treatment)
Description: The Safety Population consisted of all participants who received at least one dose of study treatment.
Arm/Group | MK-8628 Continuous Dosing Regimen 80 mg/Day | MK-8628 Continuous Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day
All-Cause Mortality (participants affected / at risk) | 3/20 | 2/4 | 1/13 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 15/20 | 3/4 | 5/13 | 3/3 | 1/6
Other Adverse Events (participants affected / at risk) | 20/20 | 4/4 | 13/13 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 Continuous Dosing Regimen 80 mg/Day (N=20) | MK-8628 Continuous Dosing Regimen 100 mg/Day (N=4) | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day (N=13) | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day (N=3) | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 Continuous Dosing Regimen 80 mg/Day (N=20) | MK-8628 Continuous Dosing Regimen 100 mg/Day (N=4) | MK-8628 Days 1-7 Dosing Regimen 100 mg/Day (N=13) | MK-8628 Days 1-7 Dosing Regimen 120 mg/Day (N=3) | MK-8628 Days 1-7 Dosing Regimen 160 mg/Day (N=6)
Anaemia (Blood and lymphatic system disorders) | 7 (19) | 2 (2) | 3 (3) | 1 (1) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Factor VII deficiency (Congenital, familial and genetic disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (10) | 1 (1) | 2 (2) | 2 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 7 (14) | 3 (5) | 6 (17)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (15) | 1 (1) | 5 (6) | 3 (10) | 5 (10)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (12) | 1 (1) | 6 (9) | 2 (3) | 3 (8)
Asthenia (General disorders) | 10 (14) | 2 (2) | 6 (8) | 0 (0) | 3 (12)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crying (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (6) | 0 (0) | 2 (3) | 2 (12) | 2 (4)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulation factor VII level increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 5 (27) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 7 (9) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 8 (13) | 1 (1) | 4 (5) | 2 (2) | 5 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (8) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subject to obligations of confidentiality, the investigator reserves the right to publish only the results of the work performed pursuant to this protocol, provided, however, that the investigator provides an authorized representative of the Sponsor with a copy of any proposed publication for review and comment at least 45 days in advance of its submission for publication.

DOCUMENTS (2):
  • Study Protocol (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02259114/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT02259114/SAP_001.pdf